CLINICAL TRIAL: NCT02789163
Title: Comparison of Diagnostic Accuracy of Automated Volume Breast Scanner to Hand Held Ultrasound for Diagnostic Breast Exam
Status: Completed | Type: Observational
Sponsor: Northeastern Ohio Radiology Research and Education Fund (Other)
Responsible Party: Principal Investigator, Richard G. Barr MD, PhD, Medical Director, Northeastern Ohio Radiology Research and Education Fund
Other Study IDs: AVBS DIAG
Record Dates: First submitted 2016-05-25; First posted 2016-06-02 (Estimated); Last update posted 2016-06-02 (Estimated); Status verified 2016-05

CONDITIONS: Breast Mass
Keywords: breast; ultrasound; diagnostic exam; automated volume breast scanner
MeSH Terms: interventions — Ultrasonography

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: Ultrasound — breast ultrasound; hand held and automated volume breast scanner

SUMMARY:
Women age >18 scheduled for a diagnostic ultrasound examination had both a hand held ultrasound and an automated breast volume scan. Exams were performed by different technologists. Images were blinded and blinded read for diagnostic accuracy of the two examinations

DETAILED DESCRIPTION:
Women aged 18 years and above presenting for a diagnostic ultrasound secondary to a palpable mass, abnormal mammogram, follow-up ultrasound abnormality, or discharge were asked to participate in the study. If the patient had both a palpable mass and a mammogram that had an abnormality the indication was listed as a palpable abnormality. Exclusion criteria included inability to give informed consent and abnormality of the breast that is larger than one quadrant. No patients were excluded from the study.

All patients received both a Hand Held (HH) and Automated Breast Volume Scanner (ABVS) ultrasound. Patients were initially randomized to have either a HH or an ABVS. The HH ultrasound was performed by one of 4 sonographers that had a minimum of 10 years experience in breast ultrasound. A different sonographer than the one performing the HH or mammography technician performed ABVS. All technologists performing ABVS participated in a training course on ABVS and performed at least 10 patients satisfactorily before beginning the study. The choice of a mammography technician or sonography to perform the ABVS was randomized. Both the sonographer performing the HH and the sonographer or mammography technologist performing the ABVS were provided the patient's history and results of the mammogram if performed for placement of the ABVS and region of interest for the HH. However the results of the HH or ABVS were not available to the person performing the second examination.

Final diagnosis was performed either by a 12 gauge core biopsy (Celero, Hologic, Marlborough, MA ) or confirmation of a benign lesion by no significant change over 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 18 years and above presenting for a diagnostic ultrasound secondary to a palpable mass, abnormal mammogram, follow-up ultrasound abnormality, or discharge were asked to participate in the study.

Exclusion Criteria:

* Unable to give informed consent
* breast abnormality greater than one quadrant

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women aged 18 years and above presenting for a diagnostic ultrasound secondary to a palpable mass, abnormal mammogram, follow-up ultrasound abnormality, or discharge were asked to participate in the study.
Sampling Method: Non-Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2013-07; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Diagnostic Accuracy | one day
  Diagnostic performance assuming BI-RADS category 1, 2, and 3 were benign and BI-RADS category 4 and 5 were malignant and using biopsy or clinical stability for two years as gold standard was assessed through ROC curves analysis. Sensitivity, specificity, Area Under the Curve (AUC) are presented along with 95% CI. Pairwise comparison of AUC between readers and methodologies are also given using z-statistics (6). P<0.05 was considered statistically significant. All tests were two-sided.

SECONDARY OUTCOMES:
Comparison of sonographer and mammography technologist performing Automated volume breast scanner | 1 day
  Diagnostic performance assuming BI-RADS category 1, 2, and 3 were benign and BI-RADS category 4 and 5 were malignant and using biopsy or clinical stability for two years as gold standard was assessed through ROC curves analysis. Sensitivity, specificity, Area Under the Curve (AUC) are presented along with 95% CI. Pairwise comparison of AUC between readers and methodologies are also given using z-statistics (6). P<0.05 was considered statistically significant. All tests were two-sided.

CONTACTS AND LOCATIONS:
Overall Officials: Richard G Barr, MD, PhD, Principal Investigator — Northeastern Ohio Radiology Research and Education Fund

IPD SHARING:
Plan to Share IPD: No